CLINICAL TRIAL: NCT05895695
Title: Levator Muscle Resection for Unilateral Congenital Ptosis Repair as Compared to Levator Plication
Brief Title: Levator Muscle Reaction for Unilateral Congenital Ptosis Repair as Compared to Levator Plication
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Maggi Hosam Wasily, resident ophthalmology department el helal hospital, Sohag University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-03-01MS
Record Dates: First submitted 2023-05-11; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Congenital Ptosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Active Comparator): evaluation of levator muscle resection on congenital ptosis
  Interventions: Procedure: levator muscle resection
- 2 (Active Comparator): evaluation of levator muscle plication on congenital ptosis
  Interventions: Procedure: levator muscle plication

INTERVENTIONS:
Procedure: levator muscle resection — resection of levator muscle in congenital unilateral ptosis
  Arms: 1
Procedure: levator muscle plication — plication of levator muscle in congenital unilateral ptosis
  Arms: 2

SUMMARY:
The aim of this study was to compare the outcome of levator muscle resection with plication in mild to moderate congenital unilateral blepharoptosis.

DETAILED DESCRIPTION:
Blepharotosis is one of the most encountered oculoplastic problems. Blepharoptosis is an abnormal low lying upper eyelid margin more than 2mm below the superior corneal limbus in the primary gaze position.

It can be subdivided according to the amount of levator function into poor (0-5),fair (6-11) or good (12 or more) millimeter. It can be classified also according to the degree of ptosis into mild (2mm) moderate (3mm) and severe ( 4mm or more). Surgical options for each of these groups are based on levator function as well as the degree and the cause of ptosis.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate simple unilateral congenital ptosis with good to fair levator function

Exclusion Criteria:

1. severe ptosis
2. poor levator function
3. poor Bell's phenomenon
4. lagophthalmos
5. diminished corneal sensation
6. completed congenital or acquired ptosis
7. history of previous lid surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Comparison of outcome of levator muscle resection and plication in mild to moderate congenital ptosis | 6 months
  Comparison of surgical efficacy of levator muscle resection and plication regarding lid height as measured by MRD 1

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] SooHoo JR, Davies BW, Allard FD, Durairaj VD. Congenital ptosis. Surv Ophthalmol. 2014 Sep-Oct;59(5):483-92. doi: 10.1016/j.survophthal.2014.01.005. Epub 2014 Feb 5. PMID 24657037
- [Background] Nemet AY. Accuracy of Marginal Reflex Distance Measurements in Eyelid Surgery. J Craniofac Surg. 2015 Oct;26(7):e569-71. doi: 10.1097/SCS.0000000000001304. PMID 26468822
- [Background] Hwang K. Surgical anatomy of the upper eyelid relating to upper blepharoplasty or blepharoptosis surgery. Anat Cell Biol. 2013 Jun;46(2):93-100. doi: 10.5115/acb.2013.46.2.93. Epub 2013 Jun 30. PMID 23869256
- [Background] Baldwin HC, Manners RM. Congenital blepharoptosis: a literature review of the histology of levator palpebrae superioris muscle. Ophthalmic Plast Reconstr Surg. 2002 Jul;18(4):301-7. doi: 10.1097/01.IOP.0000021973.72318.07. PMID 12142765